CLINICAL TRIAL: NCT05669599
Title: A Phase 2 Randomized, Placebo-controlled, Double-blind, Dose-ranging Study to Evaluate the Efficacy, Safety, and Tolerability of AMG 133 in Adult Subjects With Overweight or Obesity, With or Without Type 2 Diabetes Mellitus
Brief Title: Dose-ranging Study to Evaluate the Efficacy, Safety, and Tolerability of AMG 133 in Adult Subjects With Overweight or Obesity, With or Without Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20190218; 2023-510470-13-00 (EU CTIS Number)
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: Maridebart Cafraglutide (Experimental): Part 1: Cohort A will consist of participants without a diagnosis of type 1 or type 2 diabetes mellitus. Participants will be randomized to receive maridebart cafraglutide or placebo in 1 of 7 dose cohorts. Participants will then have the option to begin part 2 if they meet the entry criteria. Part 2: Participants that continue into part 2 will be re-randomized to receive maridebart cafraglutide or Placebo in 1 of 4 dose cohorts.
  Interventions: Biological: Maridebart Cafraglutide; Drug: Placebo
- Cohort A: Placebo (Placebo Comparator): Part 1: Cohort A will consist of participants without a diagnosis of type 1 or type 2 diabetes mellitus. Participants will be randomized to receive maridebart cafraglutide or placebo in 1 of 7 dose cohorts . Participants will then have the option to begin part 2 if they meet the entry criteria. Part 2: Participants that continue into part 2 will be re-randomized to receive maridebart cafraglutide or Placebo in 1 of 4 dose cohorts.
  Interventions: Biological: Maridebart Cafraglutide; Drug: Placebo
- Cohort B: Maridebart Cafraglutide (Experimental): Part 1: Cohort B will consist of participants with a diagnosis of type 2 diabetes mellitus. Participants will be randomized to receive maridebart cafraglutide or placebo in 1 of 4 dose cohorts. Participants will then have the option to begin part 2 if they meet the entry criteria. Part 2: Participants that continue into part 2 will be re-randomized to receive maridebart cafraglutide or Placebo in 1 of 4 dose cohorts.
  Interventions: Biological: Maridebart Cafraglutide; Drug: Placebo
- Cohort B: Placebo (Placebo Comparator): Part 1: Cohort B will consist of participants with a diagnosis of type 2 diabetes mellitus. Participants will be randomized to receive maridebart cafraglutide or placebo in 1 of 4 dose cohorts. Participants will then have the option to begin part 2 if they meet the entry criteria. Part 2: Participants that continue into part 2 will be re-randomized to receive maridebart cafraglutide or Placebo in 1 of 4 dose cohorts.
  Interventions: Biological: Maridebart Cafraglutide; Drug: Placebo

INTERVENTIONS:
Biological: Maridebart Cafraglutide — Participants will receive maridebart cafraglutide by subcutaneous (SC) injection.
  Other Names: AMG 133
Drug: Placebo — Participants will receive placebo by SC injection.

SUMMARY:
The study aims to compare and assess the dose response of 3 selected doses of maridebart cafraglutide compared with placebo, on inducing and maintaining weight loss from baseline at Week 52 in participants with overweight or obesity without diabetes mellitus (Cohort A) and in participants with overweight or obesity with Type 2 diabetes mellitus (Cohort B).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing informed consent.
* BMI ≥30 kg/m^2, or ≥27 kg/m^2 and previous diagnosis with at least one of the following comorbidities: hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease.
* For participants in cohort B only, HbA1c ≥ 7% and ≤ 10% (53 to 86 mmol/mol) at screening with an established diagnosis of type 2 diabetes mellitus for ≥ 180 days prior to screening and either treated with diet and exercise alone or on stable (at least 90 days prior to screening) treatment with metformin, a sulfonylurea, or a sodium-glucose cotransporter 2 (SGLT2) inhibitor as monotherapy or combination therapy, per approved local label.
* History of at least one unsuccessful dietary effort to lose body weight.

Exclusion Criteria:

* Change in body weight greater than 5 kg within 3 months prior to screening.
* Obesity induced by other endocrinologic disorders.
* History of pancreatitis.
* Family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2 (MEN-2).
* History of major depressive disorder within the last 2 years.
* Any lifetime history of other major psychiatric disorder or suicide attempt.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Percent Change From Baseline to Week 52 in Body Weight | Baseline and Week 52

SECONDARY OUTCOMES:
Percentage of Participants Achieving ≥ 5% Reduction in Body Weight From Baseline at Week 52 | Baseline and Week 52
Percentage of Participants Achieving ≥ 10% Reduction in Body Weight From Baseline at Week 52 | Baseline and Week 52
Achievement of ≥ 15% Reduction in Body Weight From Baseline at Week 52 | Baseline and Week 52
Achievement of ≥ 20% Reduction in Body Weight From Baseline at Week 52 | Baseline and Week 52
Change from Baseline to Week 52 in Hemoglobin A1c (HbA1c) | Baseline and Week 52
Change from Baseline to Week 52 in Fasting Serum Insulin | Baseline and Week 52
Change from Baseline to Week 52 in Fasting Plasma Glucose | Baseline and Week 52
Change from Baseline to Week 52 in Homeostasis Model Assessment for Insulin Resistance (HOMA2-IR) | Baseline and Week 52
Change from Baseline to Week 52 in Homeostasis Model Assessment for Steady State Beta Cell Function (HOMA2-%B) | Baseline and Week 52
Maximum Observed Plasma Concentration (Cmax) of maridebart cafraglutide | Up to Week 64
Area Under the Concentration-time Curve (AUC) of maridebart cafraglutide | Up to Week 64
Change from Baseline to Week 52 in Waist Circumference | Baseline and Week 52
Change from Baseline to Week 52 in Body Weight | Baseline and Week 52
Change from Baseline to Week 52 in Systolic Blood Pressure (SBP) | Baseline and Week 52
Change from Baseline to Week 52 in Diastolic Blood Pressure (DBP) | Baseline and Week 52
Change from Baseline to Week 52 in Body Fat Mass Using Dual-energy X-ray Absorptiometry (DEXA) | Baseline and Week 52
  Analyzed in a subset of participants.
Change from Baseline to Week 52 in Lean Body Mass Using DEXA | Baseline and Week 52
  Analyzed in a subset of participants.
Percent Change From Baseline to Week 52 in High-sensitivity C-reactive Protein (hs-CRP) | Baseline and Week 52
Change from Baseline to Week 52 in Body Mass Index (BMI) | Baseline and Week 52
Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) | Baseline and Week 52
Percent Change From Baseline in Total Cholesterol | Baseline and Week 52
Percent Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C) | Baseline and Week 52
Percent Change From Baseline in non-HDL-C | Baseline and Week 52
Percent Change From Baseline in Very-low-density Lipoprotein Cholesterol (VLDL-C) | Baseline and Week 52
Percent Change From Baseline in Triglycerides | Baseline and Week 52
Percent Change From Baseline in Free Fatty Acids (FFA) | Baseline and Week 52

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (78):
- United States (29):
  - Alliance for Multispecialty Research Mobile, Mobile, Alabama
  - Foothills Research Center, Phoenix, Arizona
  - HonorHealth, Scottsdale, Arizona
  - Ark Clinical Research- Long Beach, Long Beach, California
  - Ark Clinical Research- Tustin, Tustin, California
  - Orange County Research Center, Tustin, California
  - Diablo Clinical Research, Walnut Creek, California
  - Alliance for Multispecialty Research Miami, Coral Gables, Florida
  - Progressive Medical Research, Port Orange, Florida
  - East-West Medical Research, Honolulu, Hawaii
  - University of Chicago, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Alliance for Multispecialty Research Newton, Newton, Kansas
  - Louisville Metabolic and Atherosclerosis Research Center, Louisville, Kentucky
  - Tandem Clinical Research - Marrero, Marrero, Louisiana
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Alliance for Multispecialty Research Kansas City, Kansas City, Missouri
  - State University of New York Upstate Medical University, Syracuse, New York
  - Lucas Research, Morehead City, North Carolina
  - Research Innovations LLC dba Internal Medicine Care Inc, Beavercreek, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Alliance for Multispecialty Research Norman, Norman, Oklahoma
  - Medical Care LLC, Elizabethton, Tennessee
  - PanAmerican Clinical Research LLC, Brownsville, Texas
  - Headlands Research Brownsville, Brownsville, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Texas Diabetes Institute, San Antonio, Texas
- Australia (6):
  - Royal Prince Alfred Hospital (RPAH) Clinic, Camperdown, New South Wales
  - Clinical Medical and Analytical eXellence CMAX, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Heidelberg Repatriation Hospital, Heidelberg Heights, Victoria
  - Baker Heart and Diabetes Institute, Melbourne, Victoria
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - Centricity Research Brampton Endocrinology, Brampton, Ontario
  - Centricity Research Vaughan Endocrinology, Concord, Ontario
  - Institut Universitaire de cardiologie et de pneumologie de Quebec, Québec, Quebec
  - Clinique des Maladies Lipidiques de Quebec Incorporated, Québec, Quebec
- Czechia (3):
  - Endokrinologicky ustav, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut klinicke a experimentalni mediciny, Prague
- Germany (3):
  - Charite - Universitaetsmedizin Berlin, Campus Mitte, Berlin
  - Diabeteszentrum Hamburg West, Hamburg
  - Universitaetsmedizin Leipzig, Leipzig
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Hungary (4):
  - Budapesti Szent Ferenc Korhaz, Budapest
  - Clinexpert Kft, Budapest
  - CRU Hungary Kft, Encs
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Japan (9):
  - Mikannohana Clinic, Diabetes, Endocrinology and Metabolism, Matsuyama, Ehime
  - Wellness Tenjin Clinic, Fukuoka, Fukuoka
  - Matsunami Health Promotion Clinic, Hashima-gun, Gifu
  - Mazda Hospital of Mazda Motor Corporation, Aki-gun, Hiroshima
  - Nakakinen Clinic, Naka, Ibaraki
  - Nishiyamado Keiwa Hospital, Naka, Ibaraki
  - Shiraiwa Medical Clinic, Kashiwara-shi, Osaka
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - MIH Clinic Yoyogi, Shibuya-ku, Tokyo
- Poland (6):
  - AthleticoMed, Bydgoszcz
  - Centrum Badan Klinicznych PI-House Spzoo, Gdansk
  - Centrum Terapii Wspolczesnej, Lodz
  - AppleTreeClinics Network Spzoo, Lodz
  - Clinical Best Solutions Sp zoo Spolka Komandytowa, Lublin
  - Migre Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw
- South Korea (4):
  - Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kangbuk Samsung Hospital, Seoul
- Spain (4):
  - Hospital Vithas Sevilla, Castilleja de la Cuesta, Andalusia
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitario Arnau de Vilanova Lleida, Lleida, Catalonia
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Jastreboff AM, Ryan DH, Bays HE, Ebeling PR, Mackowski MG, Philipose N, Ross L, Liu Y, Burns CE, Abbasi SA, Pannacciulli N; MariTide Phase 2 Obesity Trial Investigators. Once-Monthly Maridebart Cafraglutide for the Treatment of Obesity - A Phase 2 Trial. N Engl J Med. 2025 Sep 4;393(9):843-857. doi: 10.1056/NEJMoa2504214. Epub 2025 Jun 23. PMID 40549887
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com